CLINICAL TRIAL: NCT01858961
Title: A Phase III, Randomised, Open Label, Active-controlled Study of an Interferon-free Regimen of BI 207127 in Combination With Faldaprevir and Ribavirin Compared to Telaprevir in Combination With Pegylated interferon-a and Ribavirin in Treatment-naive Patients With Chronic Genotype 1b Hepatitis C Virus Infection
Brief Title: Open Label Trial to Compare BI 207127 to Telaprevir in HCV Patients
Status: Withdrawn | Phase: Phase 3 | Type: Interventional
Sponsor: Boehringer Ingelheim (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 1241.37; 2012-004544-30 (EudraCT Number: EudraCT)
Record Dates: First submitted 2013-05-17; First posted 2013-05-21 (Estimated); Last update posted 2014-01-23 (Estimated); Status verified 2014-01

CONDITIONS: Hepatitis C, Chronic
MeSH Terms: conditions — Hepatitis C, Chronic | interventions — faldaprevir; Ribavirin; deleobuvir; telaprevir

ARMS (2):
- Group 1 (Experimental): BI 201335 in combination with BI 207127 and ribavirin for 24 weeks
  Interventions: Drug: BI 201335; Drug: ribavirin; Drug: BI 207127
- Group 2 (Experimental): Telaprevir in combination with PegIFN and ribavirin for 24 weeks or 48 weeks
  Interventions: Drug: Telaprevir; Drug: ribavirin; Drug: Pegylated Interferon

INTERVENTIONS:
Drug: BI 201335 — Once a day
  Arms: Group 1
Drug: ribavirin — Twice a day
  Arms: Group 1
Drug: BI 207127 — Twice a day
  Arms: Group 1
Drug: Telaprevir — Three times a day
  Arms: Group 2
Drug: ribavirin — Twice a day
  Arms: Group 2
Drug: Pegylated Interferon — Once a week
  Arms: Group 2

SUMMARY:
The aim of this trial is to evaluate efficacy and safety of treatment with 600 mg of BID BI 207127 in combination with 120 mg QD Faldaprevir and RBV compared to a Telaprevir-based regimen along with PegIFN and RBV in chronically infected HCV GT1 treatment naïve patients, including patients with compensated cirrhosis.

ELIGIBILITY:
Inclusion criteria:

1. Chronic HCV, diagnosed by HCV RNA = 1,000 IU/mL at screening in addition to at least one of the following:

   1. positive anti-HCV antibodies or detected HCV RNA at least 6 months prior to screening, OR
   2. liver biopsy indicating chronic HCV infection, OR
   3. history of elevated ALT levels at least 6 months prior to screening.
2. HCV infection of sub-GT1b confirmed by genotypic testing at screening.
3. Treatment naïve defined as:

   1. no prior treatment with any interferon, pegylated interferon, and /or ribavirin and
   2. no prior treatment with at least one dose of any other licensed or investigational antiviral agent for acute or chronic hepatitis C infection.
4. Availability of a liver biopsy within three years or fibroscan within 6 months prior to randomisation.

   Note: patients who do not have a liver biopsy (nor fibroscan) due to contraindication of the procedure should not be excluded for this reason. The decision on the inclusion of these patients should be discussed with the CML. Patients with a liver biopsy performed 3 or more years (or fibroscan performed 6 months or more) prior to randomisation, demonstrating cirrhosis do not need to repeat a liver biopsy or fibroscan.
5. Age 18 - 70 years (inclusive).
6. Female patients

   1. with documented hysterectomy, or
   2. who have had both ovaries removed, or
   3. with documented tubal ligation, or
   4. who are post-menopausal with last menstrual period at least 12 months prior to screening, or
   5. of childbearing potential with a negative serum pregnancy test at screening and on Day 1 (Visit 2), who agree to use two non-hormonal methods of birth control from the date of screening until 7 months after the last dose of ribavirin. They must not breast-feed at any time from the date of screening until 7 months after the last dose of ribavirin.

   Accepted methods of contraception for females in this trial are diaphragm with spermicide substances, intrauterine devices, cervical caps and condoms.

   Note: Systemic hormonal contraceptives may not be as effective in women taking BI 207127/FDV combination therapy and are not accepted methods of contraception in the study.

   OR:

   Male patients
   1. who are documented to be sterile, or
   2. who consistently and correctly use a condom while their female partners (if of child-bearing potential) agree to use one of the appropriate medically accepted methods of birth control from the date of screening until 7 months after the last dose of ribavirin, and
   3. without pregnant female partners. It is in the responsibility of the male patient to ensure that his partner (or partners) is not pregnant prior to enrolment into the study or becomes pregnant during the treatment and follow-up phase. Female partners of childbearing potential must perform monthly pregnancy tests from the date of screening until 7 months after the last dose of ribavirin (tests will be provided by the Sponsor).
7. Signed informed consent form prior to trial participation.

Exclusion criteria:

1. HCV infection of mixed genotype (1/2, 1/3, and 1/4), HCV sub-GT1a or GT1 undefined, diagnosed at screening by genotypic testing.
2. Liver disease due to causes other than chronic HCV infection which may include but is not limited to hemochromatosis, Wilson's disease, or autoimmune liver disease.
3. HIV infection.
4. Hepatitis B virus (HBV) infection based on presence of Hepatitis B surface antigen.
5. Evidence of decompensated liver disease or history of decompensated liver disease, defined as history of ascites, hepatic encephalopathy, bleeding esophageal varices or any other evidence of previous decompensation and/or any laboratory results (International Normalised Ratio, albumin, bilirubin) indicating a Child-Pugh-Turcotte score > 6 points (i.e. CPT-B or -C)
6. Confirmed or suspected active malignancy or history of malignancy within the last 5 years (with the exception of appropriately treated basal cell carcinoma of the skin or in situ carcinoma of the uterine cervix).
7. Patients with ongoing or historical photosensitivity or recurrent rash.
8. History of illicit drug use (other than cannabis) or chronic alcohol abuse within 12 months prior to randomization, in the opinion of the Investigator.
9. Body mass index <18 or >35 kg/m2.
10. Usage of any investigational drugs within 28 days prior to randomisation, or the planned usage of an investigational drug during the course of the current study.
11. Known hypersensitivity to any ingredient of the study drugs.
12. A condition that is insufficiently diagnosed, treated or clinically unstable which in the opinion of Investigator may put the patient at risk because of participation in this study, influence the results of this study, or limit the patient's ability to participate in this study.
13. Alpha fetoprotein value >100ng/mL at screening; if > 20ng/mL and = 100ng/mL, patients can be included if there is no evidence of liver cancer in an appropriate imaging study within 6 months prior to randomisation.
14. A history of severe pre-existing cardiac disease, including unstable or uncontrolled cardiac disease (e.g. congestive heart failure, myocardial infarction, unstable angina and arrhythmic disorders) current or within the previous 12 months before randomisation. Clinically significant Electrocardiogram (ECG) abnormalities. A history of congenital QT prolongation, or a family history of congenital QT prolongation or sudden death.
15. Received silymarin (milk thistle) or glycyrrhizin or Sho-saiko-to (SST) within 28 days prior to randomisation or any medication listed in a restricted medication list provided in ISF within 28 days prior to randomisation, with the exception of parenteral analgesics used during liver biopsy procedure.
16. Pre-existing psychiatric conditions that could interfere with the subject's participation in and completion of the study including but not limited to severe depression or hospitalization for depression, suicidal ideation and attempted suicide, schizophrenia, bipolar illness, severe anxiety or personality disorder, history of craniocerebral trauma or active seizure disorders requiring medication, a period of disability or impairment due to a psychiatric disease current or within the previous 3 years before randomisation.
17. Abnormal thyroid function that cannot be controlled effectively by medication.
18. Active autoimmune-mediated disease (e.g., Crohn's disease, ulcerative colitis, idiopathic thrombocytopenic purpura, systemic lupus erythematosus, autoimmune hemolytic anemia, scleroderma, severe psoriasis).
19. Requirement for chronic systemic corticosteroids (inhaled or nasally administered or pulmonary steroids will be allowed).
20. History or other evidence of severe retinopathy or clinically significant ophthalmological disorder due to diabetes mellitus or hypertension (but not limited to these conditions).

Plus other exclusion criteria relating to Peg interferon, ribavirin and Telaprevir.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2013-05; Primary Completion 2016-07 (Estimated); Study Completion 2016-07 (Estimated)

PRIMARY OUTCOMES:
Sustained Virologic Response at Week 12 after end of treatment (SVR12) | at week 12 post treatment

SECONDARY OUTCOMES:
SVR4: Plasma HCV RNA level <25 IU/mL1 at 4 weeks after end of treatment | at week 4 post treatment
SVR24: Plasma HCV RNA level <25 IU/mL1 at 24 weeks after end of treatment | at week 4 post treatment
Virological Response at Week 4 -Plasma HCV RNA level undetectable at Week 4 -Plasma HCV RNA level <25 IU/mL at Week 4 | at week 4 post treatment
Plasma HCV level undetectable at Week 12 | at week 12
Time to achieving HCV RNA undetectable | up to week 48
Virological breakthrough | up to week 48
ETR: Plasma HCV RNA level undetected at the end of treatment | week 24 or 48
Lack of on-treatment viral response | up to week 48
Relapse | up to 48 weeks post treatment
Adverse events | up to week 48 post treatment
Adverse events leading to discontinuation | up to week 48
Serious Adverse Events | up to week 48 post treatment
Laboratory test abnormalities by DAIDS grades | up to week 48 post treatment
Rate of red blood cell transfusion | up to week 48 post treatment
Time to discontinuation of trial medication | up to week 48
Liver disease progression, fibroscan and FibroSURE | up to week 48 post treatment
Rate of ESA use | up to week 48 post treatment
Change in laboratory test values over time | up to week 48 post treatment
Patients requiring hospitalisation due to AEs related to study drugs | up to week 48 post treatment

CONTACTS AND LOCATIONS:
Overall Officials: Boehringer Ingelheim, Study Chair — Boehringer Ingelheim
Locations (12):
- Australia (3):
  - 1241.37.61002 Boehringer Ingelheim Investigational Site, Westmead, New South Wales
  - 1241.37.61001 Boehringer Ingelheim Investigational Site, Adelaide, South Australia
  - 1241.37.61003 Boehringer Ingelheim Investigational Site, Fitzroy, Victoria
- Spain (7):
  - 1241.37.34010 Boehringer Ingelheim Investigational Site, Alzira
  - 1241.37.34005 Boehringer Ingelheim Investigational Site, Barcelona
  - 1241.37.34002 Boehringer Ingelheim Investigational Site, L'Hospitalet Llobregat (bcn)
  - 1241.37.34001 Boehringer Ingelheim Investigational Site, Madrid
  - 1241.37.34003 Boehringer Ingelheim Investigational Site, Madrid
  - 1241.37.34004 Boehringer Ingelheim Investigational Site, Madrid
  - 1241.37.34006 Boehringer Ingelheim Investigational Site, Valencia
- Sweden (2):
  - 1241.37.46002 Boehringer Ingelheim Investigational Site, Lund
  - 1241.37.46001 Boehringer Ingelheim Investigational Site, Stockholm